CLINICAL TRIAL: NCT01232972
Title: Oocyte Cryopreservation
Acronym: egg freezing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study technique has been declared part of standard care
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-203A
Record Dates: First submitted 2010-10-29; First posted 2010-11-02 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Fertility
Keywords: vitrification; egg freezing; oocyte cryopreservation; female fertility potential; fertility preservation; Fertility preservation, female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- oocyte freezing (Experimental): includes any women who elects to preserve her fertility by vitrifying her unfertilized eggs.
  Interventions: Procedure: vitrification of oocytes

INTERVENTIONS:
Procedure: vitrification of oocytes — eggs will be preserved via vitrification the day they are retrieved from the participant

SUMMARY:
The purpose of this investigation is to offer the opportunity for young women to cryopreserve (freeze) their oocytes (eggs) for use with IVF at a later point in time.

ELIGIBILITY:
Inclusion Criteria:

* women between the ages of 18 and 42
* election to preserve fertility by freezing eggs

Exclusion Criteria:

* women over the age of 43
* patient unwilling to sign informed consent

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2010-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Successful pregnancy | until the patient reaches 50 years of age
  Eggs will be frozen via vitrification for those females electing to preserve their fertility; patients will return following an unspecified time period, when they are ready to use their frozen eggs. At that time, the eggs will be thawed and fertilized (with the sperm source of the participant's choice) to create embryos. This time frame will be unique to each individual; however, the Center has a policy whereby no embryo transfer will be performed beyond the age of fifty (50).

SECONDARY OUTCOMES:
oocyte survival | up to 50 years of age
  the number of eggs that successfully survive the frozen-thawing procedure (vitrification).
fertilization | up to 50 years of age
  to calculate the rate for the number of oocytes that are successfully fertilized (via ICSI) following survival of the frozen-thaw procedure.
blastocyst formation | up to 50 years of age
  calculates the number of successfully fertilized embryos that grow into blastocysts (day 5 of culture), created from eggs that underwent and survived vitrification.
implantation | up to 50 years of age
  to determine the implantation rate of embryos that were created from vitrified oocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Avner Hershlag, MD, Principal Investigator — Center for Human Reproduction
Locations (1):
- Center for Human Reproduction, Manhasset, New York, United States

REFERENCES:
- [Background] Ethics Committee of the American Society for Reproductive Medicine. Fertility preservation and reproduction in cancer patients. Fertil Steril. 2005 Jun;83(6):1622-8. doi: 10.1016/j.fertnstert.2005.03.013. PMID 15950628
- [Background] Gook DA, Edgar DH. Human oocyte cryopreservation. Hum Reprod Update. 2007 Nov-Dec;13(6):591-605. doi: 10.1093/humupd/dmm028. Epub 2007 Sep 10. PMID 17846105
- [Background] Jain JK, Paulson RJ. Oocyte cryopreservation. Fertil Steril. 2006 Oct;86(4 Suppl):1037-46. doi: 10.1016/j.fertnstert.2006.07.1478. PMID 17008147
- [Background] Nagy ZP, Chang CC, Shapiro DB, Bernal DP, Kort HI, Vajta G. The efficacy and safety of human oocyte vitrification. Semin Reprod Med. 2009 Nov;27(6):450-5. doi: 10.1055/s-0029-1241054. Epub 2009 Oct 5. PMID 19806513
- [Background] Kuwayama M, Vajta G, Kato O, Leibo SP. Highly efficient vitrification method for cryopreservation of human oocytes. Reprod Biomed Online. 2005 Sep;11(3):300-8. doi: 10.1016/s1472-6483(10)60837-1. PMID 16176668
- [Background] Lee SJ, Schover LR, Partridge AH, Patrizio P, Wallace WH, Hagerty K, Beck LN, Brennan LV, Oktay K; American Society of Clinical Oncology. American Society of Clinical Oncology recommendations on fertility preservation in cancer patients. J Clin Oncol. 2006 Jun 20;24(18):2917-31. doi: 10.1200/JCO.2006.06.5888. Epub 2006 May 1. PMID 16651642
- [Background] Nagy ZP, Chang CC, Shapiro DB, Bernal DP, Elsner CW, Mitchell-Leef D, Toledo AA, Kort HI. Clinical evaluation of the efficiency of an oocyte donation program using egg cryo-banking. Fertil Steril. 2009 Aug;92(2):520-6. doi: 10.1016/j.fertnstert.2008.06.005. Epub 2008 Aug 9. PMID 18692830
- [Background] Noyes N, Boldt J, Nagy ZP. Oocyte cryopreservation: is it time to remove its experimental label? J Assist Reprod Genet. 2010 Feb;27(2-3):69-74. doi: 10.1007/s10815-009-9382-y. Epub 2010 Feb 6. PMID 20140641
- [Background] Porcu E, Venturoli S. Progress with oocyte cryopreservation. Curr Opin Obstet Gynecol. 2006 Jun;18(3):273-9. doi: 10.1097/01.gco.0000193015.96275.2d. PMID 16735826
- [Background] Nagy ZP, Diaz DG, Diaz R, Bennett A, Al-Sabagh R, V Maamari. Human oocyte preservation (Hope): preliminary results. Fertil Steril 92, Supp3:S189, 2009
- [Background] Nagy ZP, Chang CC, Bernal DP, Shapiro D, Mitchell-Leef D and Kort HI. Comparison of laboratory and clinical outcomes between fresh and vitrified sibling oocytes obtained from 30-39 year old IVF patients. Fertil Steril 92,Supp3:S67, 2009.
- [Background] Smith GD, Serafini PC, Fioravanti J, Yadid I, Coslovsky M, Hassun P, Alegretti JR, Motta EL. Prospective randomized comparison of human oocyte cryopreservation with slow-rate freezing or vitrification. Fertil Steril. 2010 Nov;94(6):2088-95. doi: 10.1016/j.fertnstert.2009.12.065. Epub 2010 Feb 19. PMID 20171613
- [Background] Practice Committees of the American Society for Reproductive Medicine and the Society for Assisted Reproductive Technology. Mature oocyte cryopreservation: a guideline. Fertil Steril. 2013 Jan;99(1):37-43. doi: 10.1016/j.fertnstert.2012.09.028. Epub 2012 Oct 22. PMID 23083924